CLINICAL TRIAL: NCT00827333
Title: Palliative Care for Quality of Life and Symptom Concerns in Family Caregivers of Lung Cancer Patients
Brief Title: Palliative Care Teaching Sessions for Family Caregivers of Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 08036; P01CA136396 (NIH); P30CA033572 (NIH); CHNMC-08036; CDR0000631261 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Early Intervention, Educational; Therapeutics; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase I-Usual Care (No Intervention)
- Phase 2 - Intervention (Active Comparator)
  Interventions: Other: educational intervention; Other: questionnaire administration; Procedure: end-of-life treatment/management; Procedure: psychosocial assessment and care; Procedure: quality-of-life assessment

INTERVENTIONS:
Other: educational intervention — Family Caregiver Palliative Care Intervention at weeks 7, 8, 10, and 12 post study enrollment
  Arms: Phase 2 - Intervention
Other: questionnaire administration — Occurs at baseline, 7 weeks, 12 weeks, 18 weeks and 24 weeks post enrollment
  Arms: Phase 2 - Intervention
Procedure: end-of-life treatment/management — Occurs at baseline, 7 weeks, 12 weeks, 18 weeks and 24 weeks post enrollment
  Arms: Phase 2 - Intervention
Procedure: psychosocial assessment and care — Occurs at baseline, 7 weeks, 12 weeks, 18 weeks and 24 weeks post enrollment
  Arms: Phase 2 - Intervention
Procedure: quality-of-life assessment — Occurs at baseline, 7 weeks, 12 weeks, 18 weeks and 24 weeks post enrollment
  Arms: Phase 2 - Intervention

SUMMARY:
RATIONALE: Palliative care teaching sessions may be more effective than standard care in improving caregiver burden, caregiver skills preparedness, quality of life, and distress in family caregivers of patients with non-small cell lung cancer.

PURPOSE: This clinical trial is studying the effects of palliative care teaching sessions in family caregivers of patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Test the effects of a family caregiver palliative care intervention (FCPCI) for informal caregivers of patients with early and late stage lung cancer on caregiver burden and caregiver skills preparedness as compared to a group of family caregivers (FC) in a usual care situation.

II. Test the effects of a FCPCI for informal caregivers of patients with early and late stage lung cancer on FC in a usual care situation.

III. Describe early and late stage FC self care behavior, comparing the usual care and FCPCI groups.

IV. Describe resource use by early and late stage FC comparing the usual care and FCPCI groups. V. Identify subgroups of FC who benefit most from the FCPCI in relation to sociodemographic characteristics, clinical/functional factors.

V. Identify subgroups of FC who benefit most from the FCPCI in relation to sociodemographic characteristics, clinical/functional factors.

OUTLINE: Family caregivers (FC) are assigned to 1 of 2 groups.

GROUP I: FC complete questionnaires at baseline and at 7, 12, 18, and 24 weeks to assess caregiver burden, caregiver skills preparedness, quality of life, distress, self care, and resource use.

GROUP II: FC undergo 4 individualized teaching sessions in weeks 7, 8, 10, and 12 that focus on caregiver burden; caregiver skills preparedness; management of patient psychological symptoms; management of FC distress; social and spiritual needs of the patient and FC; the continuing role of the FC in caring for the patient; and development of a personalized wellness plan. FC then receive 3 follow-up phone calls in weeks 16, 20, and 24 to review any questions regarding care; to assess symptom management, community resources, and support; and to review and support the wellness plan. FC also complete questionnaires as in group I.

After completion of the educational intervention, a sample of FC undergo 1-hour educational interviews exploring their perspective and insights on their experience as a caregiver.

ELIGIBILITY:
Inclusion Criteria:

* The primary family caregiver as identified by a patient with early or late stage non-small cell lung cancer (NSCLC) participating in Project 1 and 2
* Patients having been accrued to project 1 or project 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2009-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Caregiver burden | 24 weeks post study enrollment
Caregiver skills preparedness | 24 weeks post study enrollment
Caregiver quality of life | 24 weeks post study enrollment
Caregiver psychological distress | 24 weeks post study enrollment
Caregiver self-care behavior | 24 weeks post study enrollment
Resource use by caregiver | 24 weeks post study enrollment
Identification of a subgroup of caregivers who benefit most from the family caregiver palliative care intervention in relation to sociodemographic characteristics and clinical/functional factors | 24 weeks post study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Betty Ferrell, PhD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States